CLINICAL TRIAL: NCT05520684
Title: Urinary Tract Infection Risk in Women With Asymptomatic Bacteriuria or Urinalysis Abnormality at the Initiation of SGLT2 Inhibitors
Brief Title: Asymptomatic Bacteriuria, Urinalysis Abnormality at the Initiation of SGLT2 Inhibitors and UTI Risk
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Trabzon Arakli Bayram Halil Public Hospital (Other)
Responsible Party: Principal Investigator, Erman Akkus, Internal Medicine Specialist, Trabzon Arakli Bayram Halil Public Hospital
Other Study IDs: 6111449
Record Dates: First submitted 2022-08-26; First posted 2022-08-30 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Type2diabetes, SGLT2 Inhibitor, Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections | interventions — Urinalysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- positive for bacteriuria/ urinalysis abnormality: The patients who have any growth in urine culture or urinalysis abnormality at the initiation of SGLT2 inhibitor (dapagliflozin or empagliflozin)
  Interventions: Diagnostic Test: urine culture and urinalysis
- negative for bacteriuria/ urinalysis abnormality: The patients who do not have growth in urine culture or do not have abnormality in urinalysis at the initiation of SGLT2 inhibitor (dapagliflozin or empagliflozin)
  Interventions: Diagnostic Test: urine culture and urinalysis

INTERVENTIONS:
Diagnostic Test: urine culture and urinalysis — urine culture and urinalysis

SUMMARY:
The SGLT2 inhibitors have changed the treatment of type 2 diabetes mellitus in recent years, especially in patients with cardiovascular or renal disease. However, the association between SGLT2 inhibitors and urinary tract infection (UTI) risk is controversial. Moreover, it is not known whether asymptomatic bacteriuria or urinalysis abnormality at the initiation of SGLT2 inhibitors are risk factors for UTI in women. There is not enough data to recommend or not to recommend for performing urinalysis or urine culture test before initiation of SGLT2 inhibitors. The aim of the study is to investigate the effect of asymptomatic bacteriuria or urinalysis abnormality at the initiation of SGLT2 inhibitors on UTI risk in a prospective cohort of women with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Female
* >18 years old
* Type 2 Diabetes Mellitus
* Initiated SGLT2 inhibitors
* Available informed consent

Exclusion Criteria:

* Having urinary tract or genital tract symptoms at the enrollment
* Treated for urinary tract or genital tract infection in the last 3 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: The female Type 2 Diabetes Mellitus patients followed and initiated SGLT2 inhibitors by an internal medicine specialist in a public hospital covering a district
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Urinary tract infection | 3 months
  Number of participants with urinary tract infection - Any urinary tract infection treated or diagnosed by the physician clinically or by testing

CONTACTS AND LOCATIONS:
Overall Officials: Erman Akkus, MD, Study Chair — Trabzon Arakli Bayram Halil Public Hospital
Locations (1):
- Trabzon Araklı Bayram Halil Public Hospital, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No